CLINICAL TRIAL: NCT02515500
Title: Cigarette Reduction Using the Quitbit Digital Lighter and Mobile Application for Smoking Cessation: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Quitbit, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-18722
Record Dates: First submitted 2015-07-30; First posted 2015-08-04 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Smoking Cessation
Keywords: cigarette reduction; digital health; mobile health; technology; Quitbit; mHealth; smoking cessation; quit smoking; self-regulation
MeSH Terms: conditions — Smoking Cessation; Self-Control

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gradual Cessation (Active Comparator)
  Interventions: Behavioral: Gradual Cessation
- Gradual Cessation w/ Quitbit (Experimental)
  Interventions: Behavioral: Gradual Cessation w/ Quitbit

INTERVENTIONS:
Behavioral: Gradual Cessation
  Other Names: Cigarette Reduction
  Arms: Gradual Cessation
Behavioral: Gradual Cessation w/ Quitbit
  Other Names: Cigarette Reduction w/ Quitbit
  Arms: Gradual Cessation w/ Quitbit

SUMMARY:
The study is designed to evaluate the efficacy of a cigarette reduction intervention using a novel device called the Quitbit, a digital lighter paired with a smartphone mobile application, to enhance self-regulatory techniques for reducing cigarettes smoked per day toward cessation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* cigarette smoker
* wanting to quit in the next 30 days
* preference to quit gradually (vs. abruptly) or having no preference
* access to an iPhone (iOS only)
* completion of a run-in period

Exclusion Criteria:

* no major change in number of cigarettes per day in the past month (+/- 20%)
* no major health diagnoses that could impact study attrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Saliva cotinine level | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States